CLINICAL TRIAL: NCT01872728
Title: Efficacy of Facial Block for Outpatient Rhinoplasty Analgesia
Brief Title: Facial Block for Outpatient Rhinoplasty Analgesia
Acronym: FABLORA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012.774; 2012-005831-97 (EudraCT Number)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Outpatient Rhinoplasty
Keywords: facial block; levobupivacaine; regional anesthesia; rhinoplasty; outpatient

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): placebo for the realization of the facial block and morphine for intraoperative analgesia
  Interventions: Drug: Bilateral facial block after general anesthesia before surgery
- Levobupivacaine (Active Comparator): Levobupivacaine for the realization of the facial block and placebo for intraoperative analgesia
  Interventions: Drug: Bilateral facial block after general anesthesia before surgery

INTERVENTIONS:
Drug: Bilateral facial block after general anesthesia before surgery — Bilateral facial block (infraorbital and infratrochlear) after general anesthesia before surgery with intravenous placebo or bilateral block with placebo and intravenous morphine

SUMMARY:
A bilateral facial block (infraorbital and infratrochlear) will be performed immediately after intubation in patients undergoing outpatient rhinoplasty with 2.5% levobupivacaine (intervention group) or saline as control. Intravenous saline or morphine will be administered at the end of surgery in intervention or control groups, respectively. In case of pain in post-anesthesia care unit (numerical pain score >3 on a 0-10 scale), both groups will receive intravenous morphine titration. The total perioperative morphine consumption (intraoperative and in post-anesthesia care unit) will be compared between groups. Pain intensity, presence of nausea/vomiting and patient's satisfaction will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient rhinoplasty
* American Society of Anesthesiologists (ASA) classification I-II
* Affiliated to Social Security
* Written informed consent

Exclusion Criteria:

* Allergy to levobupivacaine
* Incapacity to give consent
* Chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption during the perioperative period (operating theater and post-anesthesia care unit) | J0
  At the end of post-anesthesia care unit stay

SECONDARY OUTCOMES:
Pain intensity in post-anesthesia care unit | J0 (At arrival in post-operative care unit)
  0-10 numerical rating scale (NRS) : from 0 = no pain to 10 = worst pain imaginable
Postoperative nausea and vomiting | J1 (At day 1 after surgery)
  Presence or absence of nausea/vomiting
Patient satisfaction at day 1 | J1 (At day 1 after surgery)
  0-3 scale (0 = bad, 1 = poor, 2 = good, 3 = excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France